CLINICAL TRIAL: NCT01941641
Title: A Phase II Study of Neoadjuvant FOLFOXIRI Followed by Concurrent Capecitabine and Radiotherapy for High Risk Rectal Cancer
Brief Title: Colon Neoadjuvant FOLFOXIRI Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Cancer Trials Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL021
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neoadjuvant FOLFOXIRI (Experimental)
  Interventions: Drug: neoadjuvant FOLFOXIRI; Drug: Capecitabine

INTERVENTIONS:
Drug: neoadjuvant FOLFOXIRI
Drug: Capecitabine

SUMMARY:
Objective tumour response rate to FOLFOXIRI to pre-operative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of either sex.
* ECOG performance status 0-1
* Measurable disease by RECIST 1.1 criteria.
* Histologically confirmed rectal adenocarcinoma (defined as either mid- or low rectal cancer that is located within 12 cm from the anal verge OR below the peritoneal reflection) that is previously untreated.
* 'High risk' rectal cancer, or rectal cancers that are considered marginally operable where there is a significant risk of positive surgical margin:

  * T3 (low-lying tumour at or below the levators) or T4, or
  * Tumour infiltrating perirectal fat, or
  * Any T-stage (T1-4) and node-positive tumour (invading surrounding structures or peritoneum)
* Adequate bone marrow, renal and hepatic function as defined by: absolute neutrophil count >= 1.5 x 109/L, hemoglobin >= 9 g/L, platelets >= 100 x 109/L, calculated creatinine clearance >= 55 ml/min, total bilirubin =<1.5 x the upper limit of normal, alanine aminotransferase (ALT) =<2.5 upper limit of normal.

Exclusion Criteria:

* Known distant metastasis, even if the metastasis has been resected.
* History of another invasive malignancy within the last 5 years, except for treated basal cell carcinoma of the skin, cervical intraepithelial neoplasia, or non-invasive DCIS of the breast.
* Upper rectal cancer that is located above the peritoneal reflection.
* Primary tumour associated with any one of the following features:

  * Frank intestinal obstruction, or
  * Endoscope unable to pass through the tumour's lumen plus worsening local obstructive symptoms. Note: Patients with such features should be assessed by the surgical team regarding stomal bypass prior to study enrolment. Such patients can still be considered for study enrolment after undergoing stomal bypass.
* Known hypersensitivity reaction to the study drugs (i.e. fluoropyrimidine, irinotecan, oxaliplatin)
* Known peripheral neuropathy of grade 2 or more in severity.
* Patients who have received an experimental anticancer therapy within the last 28 days.
* Previous pelvic radiotherapy. Previous oxaliplatin or irinotecan for the treatment of colon or rectal cancer
* Patient with hip prosthesis
* Major surgery within the last 28 days. Exception: Any patient who underwent stomal bypass for obstructing primary tumour within the last 14 days are still eligible, as long as the patient has sufficiently recovered from the surgery at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective tumour response rate | 2 years

SECONDARY OUTCOMES:
Tumour regression grade | 2 years
pathologic complete response | 2 years
Rate of circumferential resection margin (CRM) clearance | 2 years
Rate of tumour downstaging | 2 years
Number of Participants with Adverse Events | 2 years
Overall survival | 5 years
disease-free survival, relapse-free survival | 5 years
Time to local (and distant) recurrence | 5 years
Number of patients with 30-day post-operative mortality | 1 month
Compliance to study treatment | 2 years
Number of response to neoadjuvant therapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigette MA, MD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Hong Kong, Hong Kong